CLINICAL TRIAL: NCT05048355
Title: Metabolic Cost of Level Ground Walking With Passive vs. Powered Microprocessor Controlled Knees for Higher Active TF Amputees
Brief Title: Metabolic Cost of Walking With Passive vs. Powered Microprocessor Controlled Knees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CII2021050747
Record Dates: First submitted 2021-09-03; First posted 2021-09-17 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2021-09

CONDITIONS: Amputation; Prosthesis User
Keywords: Metabolic cost; Powered prosthetics; Microprocessor controlled knees; MPKs

STUDY DESIGN:
Intervention Model Description: single group repeated measures crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Power Knee Mainstream Dynamic (Experimental): Users are measured using their prescribed microprocessor knee and after wearing the Power Knee Mainstream dynamic for the adaptation period, they are measured again.
  Interventions: Device: Power Knee Mainstream Dynamic; Device: Passive microprocessor controlled knee

INTERVENTIONS:
Device: Power Knee Mainstream Dynamic — Powered Microprocessor controlled prosthetic knee. The Power Knee Mainstream - Dynamic, was designed to provide powered swing dynamics to restore muscle activity and thereby attempting to mitigate this increase in metabolic cost that individuals living with TF amputation face.
Device: Passive microprocessor controlled knee — Any passive microprocessor controlled prosthetic knee on the market

SUMMARY:
This study is conducted to evaluate the efficacy of the Power Knee Mainstream Dynamic compared to passive microprocessor-controlled knees (MPKs) regarding metabolic cost for high active transfemoral amputees.The test is of a single group repeated measures crossover design. The primary endpoint is the difference in MET/HRI-VO2 index between conditions. Subjects are measured on their prescribed device at visit 1, be fitted to the PKM which they wear as their primary prosthesis for one week before coming for visit 2 and being measured again on the PKM.

DETAILED DESCRIPTION:
The metabolic cost of ambulation for individuals living with a lower limb amputation is significantly increased compared to able-bodied individuals. Individuals living with transfemoral amputation have shown up to 65% more exertion to generate half the ambulation speed of able-bodied individuals.

The Power Knee Mainstream - Dynamic, was designed to provide powered swing dynamics to restore muscle activity and thereby attempting to mitigate this increase in metabolic cost that individuals living with TF amputation face. This study aims to evaluate this indirectly by measuring the heart rate during level ground walking on the Power Knee Mainstream - Dynamic compared to a passive MPK.

Previous studies reported in the literature on previous versions of the Power Knee have shown that it provides active flexion and extension during walking2, 3, 4 and more symmetric gait5 compared to passive microprocessor-controlled knees (MPKs). By providing increased symmetry and active swing during level ground walking the knee is meant to lower the effort needed by the transfemoral prosthesis user to swing the leg forward and thereby lower the metabolic cost of level ground walking.

This underpins the hypothesis being tested in this investigation, that the Power Knee Mainstream - Dynamic enables the user to walk with less metabolic cost compared to passive MPKs.

A pilot investigation that was conducted with 5 subjects indicated that the Power Knee Mainstream - Dynamic enabled users to walk on level ground with less metabolic cost compared to passive MPKs, however the difference did not reach statistical significance. The same study procedure will be used in this study with sufficient sample size to achieve the statistical power needed, which was determined in a power analysis using data form the pilot study mentioned above.

The primary objective of this study is to evaluate the efficacy of the investigational device compared to passive microprocessor-controlled knees (MPKs) regarding metabolic cost for high active transfemoral amputees.

The test is of a single group repeated measures crossover design. Amputees are a small proportion of the general population. The primary endpoint is the difference in MET/HRI-VO2 index between conditions.

Testing takes place in Össur HQ in Iceland as well as in Össur facility in Germany, the collective sample size in both sites is 20 subjects.

Subjects are measured on their prescribed device at visit 1, be fitted to the PKM which they wear as their primary prosthesis for one week before coming for visit 2 and being measured again on the PKM.

If a subject in the study is a current PKM user the procedure will apply in reverse and they will be provided with a Rheo knee to act as a comparator.

Prior to the first visit subjects will be contacted via telephone and asked screening questions, if they fit the inclusion criteria they will be booked for study visit 1. They will receive instructions to consume no alcohol and perform no exercise for 24 hours before study visit 1, the same applies to visit 2. In addition, they will be instructed to consume no caffeine prior to the visits (same day) or drink the same amount before both visits and keep the same routine the 24 hours prior to visit 1 and 2 (breakfast, water/drink consumption etc.).

During the one week follow up, subjects will be called via telephone to check the status of the device and the alignment and if there are issues identified they will be asked to come in to correct those

ELIGIBILITY:
Inclusion Criteria:

* 50Kg< body weight < 116Kg
* Cognitive ability to understand all instructions and questionnaires in the study;
* Higher active unilateral trans-femoral amputees
* Allows for 37mm knee center height to dome of pyramid alignment to allow for symmetrical knee height to sound side
* Willing and able to participate in the study and follow the protocol
* Comfortable and stable socket fit
* No socket issues/changes in the last 6 weeks
* No residual limb pain affecting functional ability
* Users with at least 6 months experience on a prosthesis

Exclusion Criteria:

* Hip disarticulation amputees
* Bilateral amputees
* Users with Osseointegrated prosthesis
* Users with co-morbidities in the contra-lateral limb, which significantly affect their functional mobility
* Users taking beta-adrenergic blocking agents (beta blockers) or other medication for heart rate control e.g. Verapamil & Digoxin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Metabolic cost | 1 week
  MET/HRI-VO2 index

CONTACTS AND LOCATIONS:
Locations (2):
- Össur Germany, Bayreuth, Bavaria, Germany
- Össur HQ, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No